CLINICAL TRIAL: NCT04179214
Title: Effects of Thoracic Spine Manipulation on Pressure Pain Sensitivity of Active Myofascial Trigger Points in Rhomboid Muscle
Brief Title: Thoracic Spine Manipulation on Pressure Pain Sensitivity of Active Myofascial Trigger Points in Rhomboid Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Bibi Haleema
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Trigger Points
Keywords: Trigger Area

STUDY DESIGN:
Intervention Model Description: Both experimental and control groups will be treated simultaneously with one treatment option common to both groups
Who Masked: Participant
Masking Description: This study will be single blinded randomized control trail, participants will be unaware of treatment groups, they will be randomly allocated through sealed envelope method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I Experimental: thoracic manipulation (Experimental): The experimental group will receive thoracic manipulation along with conventional pt protocol.
  Interventions: Other: Thoracic manipulation
- Group II Control (Active Comparator): this group of participant will receive Conventional physical therapy protocol
  Interventions: Other: conventional pt protocol

INTERVENTIONS:
Other: Thoracic manipulation — Session will be performed twice a week for a three week period if a pop sound occurred then the therapist moved on next procedure ,if not subject will be repositioned and technique will performed again. This procedure will be performed for maximum of two attempts. Approximately 3 minutes of time is required to complete thrust manipulation subjects assigned to thrust manipulation also received general exercise program and manual pressure release technique as the control group. General exercise group involve Stretching exercises for the pectoral muscles and resisted strengthening exercises for the scapular retractors and elevators and the glenohumeral abductors and external rotators were performed three times per week for 3 weeks.
  Arms: Group I Experimental: thoracic manipulation
Other: conventional pt protocol — This group will receive manual pressure release technique along with general exercises program. General exercise group involve Stretching exercises for the pectoral muscles and resisted strengthening exercises for the scapular retractors and elevators and the glenohumeral abductors and external rotators were performed three times per week for 3 weeks.
  Arms: Group II Control

SUMMARY:
This study intends to determine the effects of thoracic manipulation on pressure pain sensitivity in patients with rhomboid active trigger points.

DETAILED DESCRIPTION:
This is a single blinded controlled trial and will be conducted at physiotherapy clinic of women institute of rehabilitation sciences Abbottabad. The "screw" manipulation is a fairly aggressive manipulative technique in which the transverse processes are forced into a posterior to anterior direction Individual will be screened out according to inclusion criteria. Individuals will be allocated randomly into two groups, 30 in thoracic manipulation group and 30 in conventional physiotherapy protocol group by sealed envelope method. Both groups will receive conventional physiotherapy protocol (manual pressure release technique and muscle imbalances exercises) for rhomboid trigger points in common and the experimental group will receive thoracic manipulation in addition to conventional protocol.

Assessment will be done on baseline and after 3 weeks. Data will be analyzed on SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 30 years
* Participants presented with interscapular pain
* Forward head posture with active trigger points in rhomboid muscle
* Segmental hypomobility in upper thoracic identified with positive springing test

Exclusion Criteria:

* Participants who demonstrated contraindication to manipulation
* Open wounds or Trauma to the area which occurred less than two months prior treatment
* Any neurological compromise
* Mid scapular pain due to degenerative process or osteoporosis

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | Baseline
  Numeric pain rating scale (NPRS) is an 11 point (0-10) Scale used to measure pain. Patient verbally select value between (0-10) on the basis of intensity of pain. (0) means No pain and (10) means maximum pain experienced at baseline and after 3 weeks
Numeric pain rating scale (NPRS) | post 3 weeks
  Numeric pain rating scale (NPRS) is an 11 point (0-10) Scale used to measure pain. Patient verbally select value between (0-10) on the basis of intensity of pain. (0) means No pain and (10) means maximum pain experienced at baseline and after 3 weeks
Pain pressure threshold | baseline
  It is measured with the help of an instrument called Algometer. The readings of Algometer are both in pounds and kilograms and it gauges the pressure at which patient feels pain.
Pain pressure threshold | post 3 weeks
  It is measured with the help of an instrument called Algometer. The readings of Algometer are both in pounds and kilograms and it gauges the pressure at which patient feels pain.
Thoracic ROM | Baseline
  A thoraxic range of motion (TROM) inclinometer will be use to assess thoracic range of motion in flexion and extension.. Participants will be seated or standing upright and asked to actively move their trunk in forward and backward direction
Thoracic ROM | post 3 weeks
  A thoraxic range of motion (TROM) inclinometer will be use to assess thoracic range of motion in flexion and extension.. Participants will be seated or standing upright and asked to actively move their trunk in forward and backward direction

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | Baseline
  Neck Disability Index (NDI) is a questionnaire designed to assess how neck pain has affected patient's ability to manage in everyday life. It has total 10 sections, For each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. If all ten sections are completed the score is calculated and converted into percentages. The maximum Score of Neck Disability Index (NDI) is 50. It is measured at Baseline before Intervention and after end of treatment session that is 3 weeks
Neck Disability Index (NDI) | post 3 weeks
  Neck Disability Index (NDI) is a questionnaire designed to assess how neck pain has affected patient's ability to manage in everyday life. It has total 10 sections, For each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. If all ten sections are completed the score is calculated and converted into percentages. The maximum Score of Neck Disability Index (NDI) is 50. It is measured at Baseline before Intervention and after end of treatment session that is 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Women Institute of Rehabilitation Sciences, Abbottabad, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schiller L. Effectiveness of spinal manipulative therapy in the treatment of mechanical thoracic spine pain: a pilot randomized clinical trial. J Manipulative Physiol Ther. 2001 Jul-Aug;24(6):394-401. doi: 10.1067/mmt.2001.116420. PMID 11514816
- [Background] Ruiz-Saez M, Fernandez-de-las-Penas C, Blanco CR, Martinez-Segura R, Garcia-Leon R. Changes in pressure pain sensitivity in latent myofascial trigger points in the upper trapezius muscle after a cervical spine manipulation in pain-free subjects. J Manipulative Physiol Ther. 2007 Oct;30(8):578-83. doi: 10.1016/j.jmpt.2007.07.014. PMID 17996549
- [Background] Dunning JR, Cleland JA, Waldrop MA, Arnot CF, Young IA, Turner M, Sigurdsson G. Upper cervical and upper thoracic thrust manipulation versus nonthrust mobilization in patients with mechanical neck pain: a multicenter randomized clinical trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):5-18. doi: 10.2519/jospt.2012.3894. Epub 2011 Sep 30. PMID 21979312
- [Background] Nilsson N, Christensen HW, Hartvigsen J. The effect of spinal manipulation in the treatment of cervicogenic headache. J Manipulative Physiol Ther. 1997 Jun;20(5):326-30. PMID 9200048
- [Background] Cleland JA, Glynn P, Whitman JM, Eberhart SL, MacDonald C, Childs JD. Short-term effects of thrust versus nonthrust mobilization/manipulation directed at the thoracic spine in patients with neck pain: a randomized clinical trial. Phys Ther. 2007 Apr;87(4):431-40. doi: 10.2522/ptj.20060217. Epub 2007 Mar 6. PMID 17341509
- [Derived] Haleema B, Riaz H. Effects of thoracic spine manipulation on pressure pain sensitivity of rhomboid muscle active trigger points: A randomized controlled trial. J Pak Med Assoc. 2021 Jul;71(7):1720-1724. doi: 10.47391/JPMA.02-256. PMID 34410234